CLINICAL TRIAL: NCT01754493
Title: Open Trial of Duloxetine in Outpatients With Irritable Bowel Syndrome Symptoms and Co-Morbid Major Depression
Acronym: IBS-MDD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Roberto Lewis-Fernandez, Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #6479R; F1J-US-X037 (Other Grant/Funding Number: Eli Lilly and Company)
Record Dates: First submitted 2012-12-11; First posted 2012-12-21 (Estimated); Results first posted 2016-11-25 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Major Depression; Irritable Bowel Syndrome
Keywords: Major Depression; Irritable Bowel Syndrome; Somatization; Cymbalta; Duloxetine
MeSH Terms: conditions — Depressive Disorder, Major; Irritable Bowel Syndrome | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with Duloxetine (Experimental): Patients will receive open treatment with Duloxetine
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — This study is a 12-week open trial to assess the efficacy of duloxetine (Cymbalta) for the treatment of Irritable Bowel Syndrome (IBS) symptoms and comorbid Major Depressive Disorder (MDD). Participants will visit the clinic 8 times to meet with the psychiatrist. They will receive duloxetine to see if it helps their major depression and Irritable Bowel symptoms.
  Other Names: Cymbalta

SUMMARY:
This study will evaluate the efficacy of duloxetine in reducing depressive symptoms, abdominal pain, and other symptoms of Irritable Bowel Syndrome (IRS) in a population of outpatients with Major Depressive Disorder MDD and clinical symptoms of IBS.

DETAILED DESCRIPTION:
This study is a 12-week open trial to assess the efficacy of duloxetine (Cymbalta) for the treatment of Irritable Bowel Syndrome (IBS) symptoms and comorbid Major Depressive Disorder (MDD).

Participants will visit the clinic 8 times to meet with the psychiatrist. They will receive duloxetine to see if it helps their major depression and Irritable Bowel symptoms. Upon study completion at 12 weeks, they will receive an additional 3 months of free medication treatment at our clinic.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual,Fourth Edition (DSM-IV) criteria for major depressive disorder (MDD)
* Meets sufficient Rome III criteria for clinical symptoms of IBS
* Able to give consent
* Fluency in English or Spanish
* Patients ages 50-65 must provide a negative colonoscopy report

Exclusion Criteria:

* Current suicide risk
* History of psychosis, bipolar disorder, or a current diagnosis of Obsessive-Compulsive Disorder (OCD)
* History of alcohol or other substance abuse or dependence in the six months prior to the study
* History of non-response to an adequate trial of duloxetine
* Require concurrent treatment with other psychotropic medication or other psychiatric treatment, except zolpidem for insomnia
* Receive current treatment with a monoamine oxidase inhibitor (MAOI) within 14 days of visit 1 or potential need to use an MAOI during the study or within 5 days of discontinuation of study drug
* Patients with uncontrolled narrow-angle glaucoma
* Received electroconvulsive therapy (ECT) during the last three months
* Unable to tolerate or unwillingness to accept drug-free period of varying length: 1 week for Pro Re Nata (PRN) benzodiazepines; 2 weeks for antidepressants (other than fluoxetine), buspirone, lithium, anticonvulsants, stimulants, barbiturates, opiates, regular-use benzodiazepines (except clonazepam); 5 weeks for clonazepam and fluoxetine
* Clinically unstable medical disease including: Systemic hypertension of 140/90 mm Hg or more; known hypersensitivity to duloxetine or any of its inactive ingredients; liver function test values three times above the normal level; clinically significant thyroid dysfunction, (except patients who are stable on thyroid replacement therapy for at least three months)
* History of chronic, persisting vomiting; rectal bleeding (melena, hematochezia, Bright Red Blood Per Rectum); severe, continuous abdominal pain; nocturnal awakening with GI symptoms; weight loss not clearly related to decreased appetite of MDD; incapacitating symptoms of IBS; severe Upper GI symptoms (e.g., heartburn) that interrupt daily activities
* Family history of Ulcerative Colitis, Crohn's Disease, Celiac Disease or Colon Cancer
* Clinical findings on Physical Exam or laboratory tests of: Rectal bleeding/obstruction, elevated White Blood Cell (WBC) count, unexplained anemia, abnormal Erythrocyte Sedimentation Rate (ESR), abnormal celiac disease panel
* Evidence of clinically significant renal, pulmonary, cerebral vascular, cardiovascular, endocrine disorders, prostatic hypertrophy, urinary retention, laboratory abnormalities, abnormal electrocardiogram
* Cancer of any type. Patients in remission for 5 years or more may be judged acceptable
* Patients with current or past history of seizure disorder (except febrile seizure in childhood)
* Patients who are pregnant, breast-feeding or who do not use adequate contraceptive methods. Adequate methods include birth control pills, condom plus spermicide, an intrauterine device, the Norplant system, or diaphragm.
* Patients who are receiving effective medication for their depression or their IBS symptoms. Patients on effective medication for either disorder will be excluded.
* Patients on antidepressants and/or anti-IBS medications at intake must still meet inclusion criteria after receiving 3 months or more of medication that was dosed following FDA guidelines. Doses must have been raised so as to produce either intolerable side effects or treatment response.
* Patients who require treatment with thioridazine for any reason, at baseline and throughout the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Lewis-Fernandez, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related info — https://nyculturalcompetence.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited through print and electronic advertisements (n=12). We also received referrals from community clinicians (n=3), a former patient (n=1) and a psychiatric help line (n=1). Recruitment took place from 1/19/07 to 5/20/14.
Pre-assignment Details: This study was a single-arm open trial, so all the participants were assigned to the open-label duloxetine treatment arm.
Groups:
- Treatment With Duloxetine: Patients will receive open treatment with Duloxetine
  Duloxetine: This study is a 12-week open trial to assess the efficacy of duloxetine (Cymbalta) for the treatment of Irritable Bowel Syndrome (IBS) and comorbid Major Depressive Disorder (MDD). Participants will visit the clinic 8 times to meet with the psychiatrist. They will receive duloxetine to see if it helps their major depression and Irritable Bowel symptoms.
Period: Overall Study
Arm/Group | Treatment With Duloxetine
Started | 17
Completed | 10
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1
Not completed — Moved out of town | 1
Not completed — Scheduling conflict | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Duloxetine
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Clinician-administered 10-item scale measuring depressive symptoms (range 0-60); higher scores indicate greater severity of major depression.
Time Frame: Weeks 0, 8, 12
Population: Sample size decreased due to attrition over course of study, N=17 at Week 0, N=12 at Week 8, N=10 at Week 12. Our primary analysis was a repeated measures mixed-methods regression that included all available data points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Duloxetine
Number analyzed (Participants) | 17
units on a scale
  Week 0 | 31.59 (8.46)
  Week 8: number analyzed (Participants) | 12
  Week 8 | 15.67 (11.39)
  Week 12: number analyzed (Participants) | 10
  Week 12 | 11.4 (6.7)
Statistical Analysis 1: Comparison: Treatment With Duloxetine; We used the intention-to-treat (ITT) sample, including all subjects dispensed medication (n=17). This was a repeated-measures mixed-effects regression analysis assessing the rate of change in total MADRS symptom scores for MDD. To account for the correlation of observations within individuals, we used mixed-effects models with random intercepts and a first-order autocorrelation structure. Data from each time point (wks 0, 1, 2, 3, 4, 6, 8, 12) were used in the single repeated-measures analysis; Test type: Superiority or Other; p < .05, Mixed Models Analysis; Slope = -18.24, 95% CI 2-sided [-23.44 to -12.63]

2. Primary Outcome: Gastrointestinal Symptoms Rating Scale (GSRS)
Description: Clinician-administered 15-item scale measuring IBS symptoms (range 15-105); higher score indicates greater IBS severity.
Time Frame: Weeks 0, 8, 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Duloxetine
Number analyzed (Participants) | 17
units on a scale
  Week 0 | 54.76 (15.45)
  Week 8: number analyzed (Participants) | 12
  Week 8 | 36.33 (13.93)
  Week 12: number analyzed (Participants) | 10
  Week 12 | 31.4 (12.27)
Statistical Analysis 1: Comparison: Treatment With Duloxetine; We used the intention-to-treat (ITT) sample, including all subjects dispensed medication (n=17). This was a repeated-measures mixed-effects regression analysis assessing the rate of change in total GSRS symptom scores for IBS. To account for the correlation of observations within individuals, we used mixed-effects models with random intercepts and a first-order autocorrelation structure. Data from each time point (wks 0, 1, 2, 3, 4, 6, 8, 12) were used in the single repeated-measures analysis; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = -20.71, 95% CI 2-sided [-27.44 to -13.97]

3. Secondary Outcome: Clinician-Rated Global Impression Scales (CGI)
Description: Two clinician-administered scales measuring level of change in (1) depressive symptoms and (2) IBS symptoms, assessed separately. Range is 1-7, ranging from very much improved (1) to very much worsened (7).
Time Frame: Measured at weeks 0, 8, 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Duloxetine
Number analyzed (Participants) | 17
units on a scale
  CGI - Major Depression, Week 0 | 4.71 (0.85)
  CGI - Major Depression, Week 8: number analyzed (Participants) | 12
  CGI - Major Depression, Week 8 | 3.58 (0.67)
  CGI - Major Depression, Week 12: number analyzed (Participants) | 10
  CGI - Major Depression, Week 12 | 3 (0.94)
  CGI - IBS, Week 0 | 4.65 (0.70)
  CGI - IBS, Week 8: number analyzed (Participants) | 12
  CGI - IBS, Week 8 | 3.58 (0.67)
  CGI - IBS, Week 12: number analyzed (Participants) | 10
  CGI - IBS, Week 12 | 3 (0.94)
Statistical Analysis 1: Comparison: Treatment With Duloxetine; We used the intention-to-treat (ITT) sample, including all subjects dispensed medication (n=17). This was a repeated-measures mixed-effects regression analysis assessing the rate of change in CGI-MDD score. To account for the correlation of observations within individuals, we used mixed-effects models with random intercepts and a first-order autocorrelation structure. Data from each time point (weeks 0, 1, 2, 3, 4, 6, 8, 12) were used in the single repeated-measures analysis; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = -1.59, 95% CI 2-sided [-2.16 to -1.03]
Statistical Analysis 2: Comparison: Treatment With Duloxetine; We used the intention-to-treat (ITT) sample, including all subjects dispensed medication (n=17). This was a repeated-measures mixed-effects regression analysis assessing the rate of change in CGI-IBS score. To account for the correlation of observations within individuals, we used mixed-effects models with random intercepts and a first-order autocorrelation structure. Data from each time point (weeks 0, 1, 2, 3, 4, 6, 8, 12) were used in the single repeated-measures analysis; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = -1.55, 95% CI 2-sided [-1.99 to -1.11]

4. Secondary Outcome: Visual Analogue Scales (VAS)
Description: Five self-report 11-point Likert scales measuring pain severity in the following domains (one item each): overall pain, pain interfering with daily activities, headaches, back pain, and shoulder pain. Range is 0-10; higher scores indicate higher pain severity.
Time Frame: Measured at weeks 0, 8, 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Duloxetine
Number analyzed (Participants) | 17
units on a scale
  Overall pain, Week 0 | 5 (2.62)
  Pain interfering with daily activities, Week 0: number analyzed (Participants) | 16
  Pain interfering with daily activities, Week 0 | 4.94 (3.42)
  Headaches, Week 0 | 4.24 (2.19)
  Back pain, Week 0 | 5.47 (2.62)
  Shoulder pain, Week 0 | 5.29 (3.21)
  Overall pain, Week 8: number analyzed (Participants) | 12
  Overall pain, Week 8 | 6.08 (2.11)
  Pain interfering with daily activities, Week 8: number analyzed (Participants) | 12
  Pain interfering with daily activities, Week 8 | 6 (2.70)
  Headaches, Week 8: number analyzed (Participants) | 12
  Headaches, Week 8 | 4.5 (2.97)
  Back pain, Week 8: number analyzed (Participants) | 12
  Back pain, Week 8 | 5.58 (3)
  Shoulder pain, Week 8: number analyzed (Participants) | 12
  Shoulder pain, Week 8 | 5.17 (3.07)
  Overall pain, Week 12: number analyzed (Participants) | 10
  Overall pain, Week 12 | 4.1 (3)
  Pain interfering with daily activities, Week 12: number analyzed (Participants) | 10
  Pain interfering with daily activities, Week 12 | 4.8 (3.01)
  Headaches, Week 12: number analyzed (Participants) | 10
  Headaches, Week 12 | 3.4 (2.63)
  Back pain, Week 12: number analyzed (Participants) | 10
  Back pain, Week 12 | 4.9 (3.03)
  Shoulder pain, Week 12: number analyzed (Participants) | 10
  Shoulder pain, Week 12 | 4.7 (3.3)
Statistical Analysis 1: Comparison: Treatment With Duloxetine; We used the intention-to-treat (ITT) sample, including all subjects dispensed medication (n=17). This was a repeated-measures mixed-effects regression analysis assessing the rate of change in VAS score of overall pain. To account for the correlation of observations within individuals, we used mixed-effects models with random intercepts and a first-order autocorrelation structure. Data from each time point (weeks 0, 1, 2, 3, 4, 6, 8, 12) were used in the single repeated-measures analysis; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = -.03, 95% CI 2-sided [-1.16 to 1.10]
Statistical Analysis 2: Comparison: Treatment With Duloxetine; We used the intention-to-treat (ITT) sample with all subjects dispensed medication (n=17). This repeated-measures mixed-effects regression analysis assessed the rate of change in VAS score of pain interfering with daily activities. To account for the correlation of observations within individuals, we used mixed-effects models with random intercepts and a 1st-order autocorrelation structure. Data from each time point (wks 0, 1, 2, 3, 4, 6, 8, 12) were used in the single repeated-measures analysis; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = .47, 95% CI 2-sided [-1.07 to 2.01]
Statistical Analysis 3: Comparison: Treatment With Duloxetine; We used the intention-to-treat (ITT) sample, including all subjects dispensed medication (n=17). This was a repeated-measures mixed-effects regression analysis assessing the rate of change in VAS score of headaches. To account for the correlation of observations within individuals, we used mixed-effects models with random intercepts and a first-order autocorrelation structure. Data from each time point (weeks 0, 1, 2, 3, 4, 6, 8, 12) were used in the single repeated-measures analysis; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = -.59, 95% CI 2-sided [-2.28 to 1.10]
Statistical Analysis 4: Comparison: Treatment With Duloxetine; We used the intention-to-treat (ITT) sample, including all subjects dispensed medication (n=17). This was a repeated-measures mixed-effects regression analysis assessing the rate of change in VAS score of back pain. To account for the correlation of observations within individuals, we used mixed-effects models with random intercepts and a first-order autocorrelation structure. Data from each time point (weeks 0, 1, 2, 3, 4, 6, 8, 12) were used in the single repeated-measures analysis; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = -.35, 95% CI 2-sided [-1.56 to .87]
Statistical Analysis 5: Comparison: Treatment With Duloxetine; We used the intention-to-treat (ITT) sample, including all subjects dispensed medication (n=17). This was a repeated-measures mixed-effects regression analysis assessing the rate of change in VAS score of shoulder pain. To account for the correlation of observations within individuals, we used mixed-effects models with random intercepts and a first-order autocorrelation structure. Data from each time point (weeks 0, 1, 2, 3, 4, 6, 8, 12) were used in the single repeated-measures analysis; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = -.48, 95% CI 2-sided [-2.00 to 1.03]

5. Secondary Outcome: Somatization Module of the Patient's Health Questionnaire (PHQ-15)
Description: Self-report 15-item scale measuring somatization symptoms (range 0-30); higher score indicates greater severity of somatization symptoms.
Time Frame: Measured at weeks 0, 8, 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Duloxetine
Number analyzed (Participants) | 17
units on a scale
  Week 0 | 16.06 (3.75)
  Week 8: number analyzed (Participants) | 12
  Week 8 | 12.87 (4.26)
  Week 12: number analyzed (Participants) | 10
  Week 12 | 11.1 (6)
Statistical Analysis 1: Comparison: Treatment With Duloxetine; We used the intention-to-treat (ITT) sample with all subjects dispensed medication (n=17). This was a repeated-measures mixed-effects regression analysis assessing the rate of change in PHQ-15 scores of somatization symptoms. To account for the correlation of observations within individuals, we used mixed-effects models with random intercepts and a first-order autocorrelation structure. Data from each time point (weeks 0, 1, 2, 3, 4, 6, 8, 12) were used in the single repeated-measures analysis; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = -4.38, 95% CI 2-sided [-7.39 to -1.36]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The treating psychiatrist assessed adverse effects systematically at each visit by evaluating 28 potential effects with the Treatment Emergent Side Effect Scale (TESS) on a 4-point Likert scale ranging from 0 (absent) to 3 (severe).
Arm/Group | Treatment With Duloxetine
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 6/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Duloxetine (N=17)
Neck stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) — Two patients reported neck stiffness
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 2 (2) — Two patients reported muscle rigidity
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) — One patient reported nausea and vomiting
Constipation (Gastrointestinal disorders) | 1 (1) — One patient reported constipation
Sweating (General disorders) | 1 (1) — One patient reported sweating
Tachycardia (Cardiac disorders) | 1 (1) — One patient reported tachycardia

LIMITATIONS AND CAVEATS:
Study limitations include the lack of placebo control, modest sample size, single ethnic group, and high attrition rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No